CLINICAL TRIAL: NCT04101630
Title: Activity Monitoring in Pulmonary Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Evan Brittain, Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: Physical Activity in PH
Record Dates: First submitted 2019-09-16; First posted 2019-09-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with Pulmonary Hypertension: Participants will undergo activity monitoring for 12 weeks, at baseline and once a year for 3 years. Patient reported outcomes will be collected including Quality of Life questionnaires [emphasis-10, Minnesota Living with Heart Failure (MLHF), and SF-36 surveys], medication changes, hospitalization, and death.
  Interventions: Behavioral: Activity Monitoring
- Healthy Volunteers: Participants will undergo activity monitoring for 12 weeks, at baseline and once a year for 3 years. Patient reported outcomes will be collected including Quality of Life questionnaires [emphasis-10, Minnesota Living with Heart Failure (MLHF), and SF-36 surveys], medication changes, hospitalization, and death.
  Interventions: Behavioral: Activity Monitoring

INTERVENTIONS:
Behavioral: Activity Monitoring — Monitoring with FitBit

SUMMARY:
This is a prospective, longitudinal, observational study of free-living activity trackers and patient reported outcomes to test the hypothesis that daily activity will have stronger prognostic value than 6MWD in patients with pulmonary hypertension after 12 weeks.

DETAILED DESCRIPTION:
A prospective, longitudinal, observational study of free-living activity tracking and patient-reported outcomes in patients with pulmonary hypertension. Participants will undergo activity monitoring for 12 weeks once a year for 4 years. Patient-reported outcomes will be collected including quality of life (emphasis-10, Minnesota Living with Heart Failure (MLHF), and SF-36 surveys), medication changes, hospitalization, and death. This study aims to enroll 500 participants. The objectives of this study are to establish the clinical utility of daily activity tracking in patients with pulmonary hypertension and to identify clinical factors associated with reduced daily activity.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in L-PVDOMICS or
* Any patient in the United States with pulmonary hypertension confirmed by hemodynamics and expert clinical diagnosis

Exclusion Criteria:

* Pregnancy
* Hospitalization within the prior 3 months
* Orthopedic limitations that preclude 6MWD testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be those enrolled in the Longitudinal Pulmonary Vascular Disease Phenomics Program (L-PVDOMICS) and any patient with pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Activity Monitoring | Baseline
  Participants will wear an accelerometer to record activity level
Activity Monitoring | 1 year
  Participants will wear an accelerometer to record activity level
Activity Monitoring | 2 year
  Participants will wear an accelerometer to record activity level
Activity Monitoring | 3 year
  Participants will wear an accelerometer to record activity level

SECONDARY OUTCOMES:
Six Minute Walk Distance (6MWD) Test | Baseline, 1 year, 2 year, 3 year
  Six Minute Walk Distance Test
Intensity of Activity | Baseline, 1 year, 2 year, 3 year
  Intensity of activity is categorized as rest, light, moderate, and vigorous based on calculated metabolic equivalents.
Quality of Life 36-Item Short Form Survey (SF-36) | Baseline, 1 year, 2 year, 3 year
  Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
emPHasis-10 | Baseline, 1 year, 2 year, 3 year
  The emPHasis-10 is a pulmonary hypertension-specific questionnaire to assess health related quality of life. It covers breathlessness, fatigue and lack of energy, social restrictions, and concerns regarding effects on patient's significant others, such as family and friends. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicating worse quality of life.
Minnesota Living with Heart Failure (MLHF) | Baseline, 1 year, 2 year, 3 year
  The MLHFQ is one of the most widely used health-related quality of life questionnaires for patients with heart failure. It provides scores for two dimensions, physical and emotional, and a total score. It is a reliable and valid patient-oriented measure of the adverse effects of heart failure on a patient's life. The score can range from 0-126 with 0 being minimal impact and 126 being high impact.

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Brittain, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Use of study data and biospecimens, and resulting findings, during the PVDOMICS study are subject to approval of the PVDOMICS Steering Committee and follow guidelines of the Publications and Ancillary Study Committee. The data and biospecimens from subjects at a clinical center are the property of the PVDOMICS study and are under the custody of that center.
  At the end of the PVDOMICS study and this proposal, the data and remaining biospecimens will be transferred to PVDOMICS and/or to the National Heart, Lung and Blood Institute (NHLBI) Biological Specimen and Data Repository Information Coordinating Center (BioLINCC) biobank and become the property of one of these organizations. Future researchers may request data or biospecimens from a biobank with approval following the guidelines of the biobank. Protocols for data sharing after the conclusion of PVDOMICS have not been established, but will be created in accordance with the NIH Data Sharing Policy.
Time Frame: at the end of the PVDOMICS study
Access Criteria: subject to approval of PVDOMICS Steering Committee